CLINICAL TRIAL: NCT03486067
Title: A Phase 1, Open-label, Dose Finding Study of CC-93269, a BCMA x CD3 T Cell Engaging Antibody, in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Study of CC-93269, a BCMA x CD3 T Cell Engaging Antibody, in Participants With Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-93269-MM-001; U1111-1210-6325 (Registry Identifier: WHO); 2023-506564-14 (Other: EU CTR)
Record Dates: First submitted 2018-03-21; First posted 2018-04-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; BCMA X CD3 T Cell; Antibody; CC-93269; Relapsed and Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-93269 (Experimental)
  Interventions: Drug: CC-93269

INTERVENTIONS:
Drug: CC-93269 — Specified dose on specified days
  Other Names: Alnuctamab

SUMMARY:
Study CC-93269-MM-001 is an open-label, Phase 1, dose escalation (Part A and C) and expansion (Parts B and D), first-in-human clinical study of CC-93269 in subjects with relapsed and refractory multiple myeloma.

DETAILED DESCRIPTION:
The dose escalation parts (Part A with CC-93269 administered intravenous (IV) and Part C subcutaneous (SC)) of the study will evaluate the safety and tolerability of escalating doses of CC-93269, administered IV or SC, to determine the maximum tolerated dose (MTD) and non-tolerated dose (NTD) of CC-93269. The expansion parts (Part B and D) will further evaluate the safety and efficacy of CC-93269 administered IV or SC at or below the MTD in selected expansion cohorts of up to approximately 20 evaluable subjects each in order to determine the Recommended Phase 2 dose (RP2D).One or more dosing regimens may be selected for cohort expansion. All treatments will be administered in 28-day cycles for up to 5 years for subjects maintaining clinical benefit, or until confirmed disease progression, unacceptable toxicity, or subject/investigator decision to withdraw.

ELIGIBILITY:
Inclusion Criteria:

* History of multiple myeloma with relapsed and refractory disease
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Must have measurable disease as determined by the central laboratory

Exclusion Criteria:

* Symptomatic central nervous system involvement of multiple myeloma
* Prior autologous stem cell transplant ≤ 3 months prior
* Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤ 12 months prior
* History of concurrent second cancers requiring active, ongoing systemic treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 63 months
  Number of participants with Adverse Events
Dose Limiting Toxicity (DLT) | Up to 60 months
  Is defined as any of the toxicities occurring within the DLT assessment window (Cycle 1, Days 1 to 28) except those that are clearly and incontrovertibly due to extraneous causes.
Non-Tolerated Dose (NTD) | Up to 60 months
  Is defined as a dose level at which 2 or more of up to 6 evaluable subjects in any dose cohort experience a DLT in the DLT window.
Maximum Tolerated Dose (MTD) | Up to 60 months
  Is defined as the last dose cohort below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during the DLT window.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 60 months
  Is defined as the proportion of subjects who achieve a partial response or better (eg, PR, VGPR, CR or sCR), according to International Myeloma Working Group (IMWG) response criteria.
Time to Response | Up to 60 months
  Is defined as the time from the first CC-93269 dose date to the date of first documented response (PR or better).
Duration of Response | Up to 60 months
  Is defined as the time from the earliest date of documented response (≥ PR) to the first documented disease progression or death, whichever occurs first.
Progression Free Survival | Up to 60 months
  Is defined as the time from the first dose of CC-93269 to progressive disease or death from any cause, whichever occurs first.
Overall Survival | Up to 60 months
  Is defined as the time from the first dose of CC-93269 to death from any cause.
Pharmacokinetics - Cmax | Up to 60 months
  Maximum serum concentration of drug
Pharmacokinetics - Cmin | Up to 60 months
  Minimum serum concentration of drug
Pharmacokinetics - AUC | Up to 60 months
  Area under the curve
Pharmacokinetics - tmax | Up to 60 months
  Time to peak (maximum) serum concentration
Pharmacokinetics - t1/2 | Up to 60 months
  Terminal Half-life
Pharmacokinetics - CL | Up to 60 months
  Apparent total body clearance
Pharmacokinetics - Vss | Up to 60 months
  Volume of distribution at steady-state
Pharmacokinetics - accumulation index of alnuctamab | Up to 60 months
  Accumulation ratio of drug
Presence and frequency of anti-drug antibodies (ADA) | Up to 60 months
  Detection of anti-drug antibodies in participants and frequency of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (34):
- United States (9):
  - Local Institution - 105, Birmingham, Alabama
  - Local Institution - 103, San Francisco, California
  - Local Institution - 107, New Haven, Connecticut
  - Local Institution - 106, Atlanta, Georgia
  - Local Institution - 109, Boston, Massachusetts
  - Local Institution - 111, Boston, Massachusetts
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai Mount Sinai West, New York, New York
  - Local Institution - 101, Seattle, Washington
- Germany (5):
  - Local Institution - 305, Erlangen
  - Local Institution - 303, Hamburg
  - Local Institution - 302, Heidelberg
  - Local Institution - 306, München
  - Local Institution - 304, Tübingen
- Italy (3):
  - Local Institution - 402, Bergamo
  - Local Institution - 403, Meldola
  - Local Institution - 401, Milan
- Japan (5):
  - Local Institution - 602, Nagoya, Aichi-ken
  - Local Institution - 603, Shibuya-ku, Tokyo
  - Local Institution - 605, Kamakura
  - Local Institution - 604, Kashiwa
  - Local Institution - 601, Kyoto
- Spain (8):
  - Local Institution - 206, Barcelona
  - Local Institution - 208, Barcelona
  - Local Institution - 205, Madrid
  - Local Institution - 201, Pamplona
  - Local Institution - 203, Salamanca
  - Local Institution - 204, Santander
  - Local Institution - 207, Valencia
  - Local Institution - 202, Valencia
- Sweden (4):
  - Local Institution - 504, Gothenborg
  - Local Institution - 502, Lund
  - Local Institution - 501, Stockholm
  - Local Institution - 505, Uppsala

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com